CLINICAL TRIAL: NCT07265375
Title: Second Chance Stipends Randomized Controlled Trial
Brief Title: Second Chance Stipends RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11235
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Poverty; Incarceration
Keywords: cash transfer; incarceration; recidivism
MeSH Terms: conditions — Recidivism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Recipients of stipend
  Interventions: Other: Cash transfer
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Cash transfer — Provision on monthly cash transfer
  Arms: Treatment

SUMMARY:
Investigators will execute a mixed methods randomized controlled trial to determine the impacts of cash transfers of $750 per month for 12 months. Investigators will measure the impacts of the cash transfers on physical and mental health, housing stability, healthcare utilization, financial stability, and interactions with the criminal legal system.

DETAILED DESCRIPTION:
The transition from incarceration to community reintegration represents a finite time period of unique challenges, often exacerbated by fines and other structural constraints associated with limited access to housing, the workforce, and public benefits. As such, individuals exiting prisons are most vulnerable for recidivism and other poor wellbeing outcomes during the initial period after their release.

The project will enroll approximately 200 individuals in the Omaha, NE area to receive $750 per month over a one-year period. Another 250 will be assigned to the control group and will not receive the cash transfers but will be eligible to participate in research activities. Adults exiting Nebraska state prisons will be eligible to participate if they are exiting prison during the specified time frame and do not have a conviction of a sex crime or homicide.

Longitudinal repeated measures will be utilized through surveys conducted at baseline, 6 months, 12 months, and 18 month intervals. Future involvement with the criminal legal system will be measured using linked administrative data from the Department of Corrections. A select group of 30 participants across study groups will also be invited to participate in in-depth interviews with a CGIR research scientist and team at multiple time points.

ELIGIBILITY:
Inclusion criteria:

* Aged 18 or older
* Exiting Nebraska state prisons during the study enrollment period

Exclusion criteria:

- Conviction of a sex crime or homicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Recidivism | 1 year following release date
  As applied to adults, recidivism shall mean a final conviction of a Class I or II misdemeanor, a Class IV felony or above, or a Class W misdemeanor based on a violation of state law or an ordinance of any city or village enacted in conformance with state law, within 1 year of being successfully released.
Post-release compliance with payment of fees | 1 year post release date or for the duration of required supervision, whichever is sooner
  Compliance/non-compliance with post-release payment of fees. A count of fee payments (continuous) and on-time payment as a binary outcome variable (y/n) for each instance.
Post-release compliance with probation officer meetings | 1 year post release date or for the duration of required supervision, whichever is sooner
  Compliance/non-compliance with post-release attendance of meetings with probation officer. A count of meetings (continuous) and attendance at meetings (y/n) for each instance.

SECONDARY OUTCOMES:
Housing status | Baseline, 6 months, 12 months
  Housing status (e.g., renter, homeowner, rent-to-own, etc.) reported in the prior month.
Food security (Household Food Insecurity Access Scale) | Baseline, 6 months, 12 months
  9 items to assess past four week food insecurity: 1) worry about not having enough food, 2) inability to eat preferred foods, 3) eating a limited variety of foods, 4) having to eat foods that they did not want to eat, 5) eating a smaller meal than needed, 6) eating fewer meals in a day, 7) having no food to eat, 8) going to sleep at night hungry, and 9) going a whole day and night without eating. Items scored as "yes" (1) or "no" (0).
Employment | Baseline, 6 months, 12 months
  Employment status as measured by one item with attributes per the U.S. Department of Labor.
Financial wellbeing (Consumer Financial Protection Bureau Financial Wellbeing Scale) | Baseline, 6 months, 12 months
  Each item is scored 0 to 4 and summed to a total. The sum total is then converted to a total response value on the CFPB Financial Well-Being Scale score from 0-100, where higher scores indicate a greater sense of financial well-being.
Psychological distress (Kessler 6) | Baseline, 6 months, 12 months
  Each item is scored from zero "none of the time" to four "all of the time." Scores of the 6 items are then summed, yielding a minimum score of 0 and a maximum score of 24. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
General health | Baseline, 6 months, 12 months
  Self-reported general health as measured by one question from the SF-36: "In general, would you say your health is:", with a 5-point scale from Poor to Excellent.
Substance use (UNCOPE) | Baseline, 6 months, 12 months
  Six items, each scored 0 (no) or 1 (yes). A score of two or more indicates possible substance misuse.

CONTACTS AND LOCATIONS:
Overall Officials: Stacia West, PhD, Principal Investigator — The University of Pennsylvania; Amy Castro, PhD, Principal Investigator — The University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No